CLINICAL TRIAL: NCT04275141
Title: Genetic Analysis Coupled to Application of Isotopic Techniques to the Study of Mauriac Syndrome
Brief Title: Mauriac Syndrome: Isotopic Techniques and Genetic Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christel Tran, Principal Investigator, University of Lausanne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NCT2019-01755
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Short Stature; Glycogen Deposition
MeSH Terms: conditions — Diabetes Mellitus; Dwarfism | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Case control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mauriac syndrome (Other): An oral dose of glucose (labelled with 1% U-13C6-glucose) will be given at time 0 min followed by a 30-min cycling exercise at time 300 min.
  Interventions: Other: oral glucose load; Other: exercise test
- Type 1 diabetes mellitus (Other): An oral dose of glucose (labelled with 1% U-13C6-glucose) will be given at time 0 min followed by a 30-min cycling exercise at time 300 min.
  Interventions: Other: oral glucose load; Other: exercise test

INTERVENTIONS:
Other: oral glucose load — oral glucose load (60g) followed by exercise at fixed wattage (60W) for 30 min
Other: exercise test — oral glucose load (60g) followed by exercise at fixed wattage (60W) for 30 min

SUMMARY:
Mauriac syndrome (MS) is an entity of individuals combining poorly controlled diabetes mellitus type 1, short stature and glycogenic hepatopathy. Thus, the functional significance of Mauriac syndrome for glucose metabolism remains disputed, and whether genetic defects in glycogen metabolism contribute to glycogenic hepatopathy in MS remains to be clarified.Coupling the genetic analysis of targeted genes involved in glucose regulation with a dynamic exploration will eventually determine if a genetic abnormality leads to the disease and explains the nature of the phenotype.

DETAILED DESCRIPTION:
Investigation of glucose homeostasis in MS, after an oral glucose load followed by exercise, using a quantitative measurement of the substrate flux. This dynamic in vivo kinetics can be explored using stable, nonradioactive tracers with the help of gas or liquid chromatography.

Investigation of genetic factors associated with MS phenotype. Molecular analysis will be performed by next generation sequencing (exome or whole genome sequencing). In addition, a targeted analysis for pathogenic variants in genes implicated in homeostasis regulation will be done.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for controls:
* DT1
* > 18 years old)
* Presence of at least one of the following auto-antibodies: anti-GAD65, anti-IAA, anti-ZnT8, anti-IA2 or ICA and/or low C-Peptide
* Insulin therapy by multiple daily injections or continuous subcutaneous insulin infusion by an insulin pump
* Informed consent as documented by signature

Inclusion criteria for subjects:

* Mauriac syndrome
* DT1
* > 18 years old
* Presence of hepatomegaly in infancy (confirmed ≥ 1 abdominal US) at the time of diagnosis of Mauriac Syndrome
* Presence of short stature during infancy at the time of diagnosis of Mauriac Syndrome (<P3; WHO growth curves on ≥ 2 different measures, at 2 different time-points)
* Presence of at least one of the following auto-antibodies: anti-GAD65, anti-IAA, anti-ZnT8, anti-IA2 or ICA and/or low C-Peptide
* Informed consent as documented by signature

Exclusion criteria for subjects and controls :

* Obesity (BMI ≥ 30 kg/m2 or > 90th percentile)
* Illness that contraindicates physical activity
* Women who are pregnant or breast feeding
* Any clinically unstable disease
* Myocardial infarcts, syncope, heart rhythm disorder, unstable hypertension in the last 6 months
* Blood donation in the last 3 months for men and 4 months for women before the study
* Enrollment in a previous study less than 30 days before the start of the study
* Participation of the investigator, a family member, an employee or someone having a link with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
In vivo kinetics of ingested glucose | Time -90 minutes to Time 360 minutes
  Plasma glucose kinetics [Time -90 min before ingestion of a test meal to Time 360 min after ingestion of a test meal]
  * Baseline : [Time -90min to Time 0min]
  * After an oral glucose load (60g): [Time 0min to Time 300min]
  * During exercise at fixed wattage (60W) for 30 min: [Time 300 min to Time 330 min]
  * After exercise for 30 min [Time 330 min to Time 360 min]
  Trial stable isotope tracers ([U-13C6] glucose ingestion, will be used to assess ingested glucose flux at baseline and during the test.
In vivo kinetics of endogenous glucose | Time -90 minutes to Time 360 minutes
  Plasma glucose kinetics [Time -90 min before ingestion of a test meal to Time 360 min after ingestion of a test meal]
  * Baseline : [Time -90min to Time 0min]
  * After an oral glucose load (60g): [Time 0min to Time 300min]
  * During exercise at fixed wattage (60W) for 30 min: [Time 300 min to Time 330 min]
  * After exercise for 30 min [Time 330 min to Time 360 min]
  Trial stable isotope tracers [6,6-2H2] glucose infusion will be used to assess endogenous glucose flux at baseline and during the test.
In vivo kinetics of lactate | Time -90 minutes to Time 360 minutes
  Plasma lactate kinetics [Time -90 min before ingestion of a test meal to Time 360 min after ingestion of a test meal]
  * Baseline : [Time -90min to Time 0min]
  * After an oral glucose load (60g): [Time 0min to Time 300min]
  * During exercise at fixed wattage (60W) for 30 min: [Time 300 min to Time 330 min]
  * After exercise for 30 min [Time 330 min to Time 360 min]
  Trial stable isotope tracers [1-13C1]lactate infusion will be used to assess lactate flux at baseline and during the test.

SECONDARY OUTCOMES:
DNA Banking | At inclusion period
  10 ml of whole blood will be collected, at baseline, in two tubes EDTA 5ml for DNA extraction and banking in view of next generation sequencing (NGS) analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Lausanne University Hospitals, Lausanne, Canton of Vaud
  - Geneva University Hospital, Geneva